CLINICAL TRIAL: NCT00553683
Title: Phase I/II Study of Autologous Tumor Cell Vaccination Using Metronomic Cyclophosphamide, 3-Dimensional Conformal Radiotherapy, Intra/Peri-Tumor Injection of Poly ICLC With Trans-Hepatic Arterial Embolization Followed by Poly ICLC Boosting in Patients With Unresectable, Recurrent, or Metastatic Cancers in the Liver (Hepatoma, Cholangiocarcinoma, Neuroendocrine, Breast, Colon, Gastric, and Esophageal Cancer)
Brief Title: Cyclophosphamide, Radiation Therapy, and Poly ICLC in Treating Patients With Unresectable, Recurrent, Primary, or Metastatic Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrew de la Torre, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000573370; UMDNJ-0120070076
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Gastric Cancer; Liver Cancer; Melanoma (Skin); Metastatic Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: stage IV pancreatic cancer; adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent pancreatic cancer; recurrent colon cancer; recurrent breast cancer; recurrent gastric cancer; recurrent ovarian epithelial cancer; recurrent melanoma; stage IV breast cancer; stage IV gastric cancer; stage IV colon cancer; stage IV ovarian epithelial cancer; stage IV melanoma; liver metastases
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Melanoma; Neoplasm Metastasis; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular; Colonic Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cyclophosphamide; poly ICLC; Radiotherapy, Conformal

ARMS (1):
- poly ICLC (Experimental)
  Interventions: Drug: cyclophosphamide; Drug: poly ICLC; Procedure: hepatic artery embolization; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: poly ICLC
Procedure: hepatic artery embolization
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Poly ICLC may stop the growth of liver cancer by blocking blood flow to the tumor. Giving the drug directly into the arteries around the tumor may kill more tumor cells. Giving cyclophosphamide and radiation therapy together with poly ICLC may be an effective treatment for liver cancer.

PURPOSE: This phase I/II trial is studying the side effects of giving cyclophosphamide, radiation therapy, and poly ICLC together and to see how well they work in treating patients with unresectable, recurrent, primary, or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To study the safety and effectiveness of a strategy to establish robust anticancer immunologic body defenses by using low-dose radiation therapy to the liver cancer in order to increase tumor targetability; inject a body defense activator, polyinosinic-polycytidylic acid polylysine carboxymethylcellulose (poly ICLC, hiltonol, oncovir), into and around the cancer to activate sentinel dendritic cells to alarm body defenses; and shut down local production of factors that suppress the body's natural anticancer defenses by starving the cancer of its blood supply within the liver.

OUTLINE: Patients receive low-dose oral cyclophosphamide once daily on days 1-21 and undergo 3-dimensional conformal radiotherapy on days 21-23. On day 24, patients undergo an intra- or peri-tumoral polyinosinic-polycytidylic acid polylysine carboxymethylcellulose (poly ICLC) injection directly into the tumor followed by trans-hepatic artery embolization to the designated tumor. Patients receive poly ICLC subcutaneously on days 26, 35, 37, 42, 44, 49, and 51. Treatment repeats every 57 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologically or histologically confirmed hepatocellular carcinoma

  * Stage III or IV primary disease
  * Recurrent, unresectable, or metastatic disease meeting any of the following criteria:

    * Pancreatic cancer that underwent prior surgical resection and progressed with recurrent metastatic disease to the liver
    * Gastric, colon, breast, or ovarian cancer or melanoma with metastatic disease to the liver
    * Primary or recurrent disease that cannot be surgically resected leaving the patient disease-free
* Radiologically measurable disease
* Ineligible for liver transplantation according to University of San Francisco listing criteria:

  * Single lesion > 6.5 cm
  * Three or more tumors > 4.5 cm
  * Cumulative tumor diameter > 8 cm

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* ANC ≥ 1,500/mm³
* Platelets ≥ 75,000/mm³
* Creatinine ≤ 1.7 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 3 times the upper limit of normal
* INR < 1.5
* LVEF ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious concurrent infection or medical illness that would render the protocol treatment unsafe
* LVEF ≥ 50%

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Overall tolerability | up to 90 days

SECONDARY OUTCOMES:
Progression-free survival at 6, 12, and 24 months | up to 24 months
Overall survival at 6, 12, and 24 months | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N. de la Torre, MD, Study Chair — UMDNJ University Hospital / St Joseph Medical Center
Locations (1):
- Rutgrers University Hospital, Newark, New Jersey, United States